CLINICAL TRIAL: NCT00186706
Title: The Effect of Selenium Supplementation on Anti-Oxidant Levels in COPD Patients: A 12-Week, Randomized, Placebo-Controlled Trial
Brief Title: Selenium Supplementation in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Health Care London (Other)
Collaborators: Father Sean O'Sullivan Research Centre (Unknown)
Organization: St. Joseph's Healthcare Hamilton (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R.P. #04-2326
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Cardiovascular Disease
Keywords: Selenium; Chronic Obstructive Pulmonaary Disease; Cardiovascular Disease; Anti-oxidant; Pulmonary
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Selenium

SUMMARY:
Does an oral selenium supplement increase blood levels of antioxidants in patients with established, smoking-related lung disease?

Members of our study group recently discovered that elevated levels of the anti-oxidant GPx-1 may be protective against heart disease. We are studying whether selenium supplementation will improve GPx-1 levels.

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) are at high risk for atherosclerotic heart disease, in part because of their nearly universal exposure to heavy smoking, and in part to other incompletely understood mechanisms which may include inflammation and anti-oxidant status.

Smoking markedly affects both circulating inflammatory markers concentrations, and the anti-oxidant glutathione peroxidase-1 (GPx-1). We hypothesize that smoking-related inflammation and anti-oxidant consumption lead to both cardiovascular (CV) and respiratory disease. In a recent study, we (Blankenberg et al) found that higher levels of GPx-1 were associated with lower rates af future CV events and death. GPx-1 levels were lower among smokers, and the combination of current smoking and GPx-1 levels below the median was strongly (HR=5.6) and significantly associated with future CV events and death.

There is a biological and epidemiological rationale to study selenium supplementation for CV protection. GPx-1 is a selenium-dependent enzyme, and data support the hypothesis that selenium supplementation increases GPx activity in various diseases. Furthermore, epidemiologic studies have discovered an inverse association between selenium content in soil and CV incidence and mortality. We hypothesize that selenium supplementation will elevate intra-erythrocytic GPx-1 levels in COPD patients and, ultimately, retard CV progression.

In this study, we will test the first component of this assertion. In a randomized, placebo-controlled trial, we will determine whether 12 weeks of selenium supplementation increases GPx-1 levels among 120 COPD patients. If successful, this study may lead to future large clinical trials to assess whether selenium, an inexpensive and safe mineral, improves clinical outcomes in cardiovascular and respiratory disease.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40 years or older (no upper limit).
2. Established Respirologist-diagnosed mild or moderate COPD, according to the Canadian Thoracic Society (CTS) Lung Function Guidelines.(33) For a diagnosis of mild COPD, patients must have FEV1 60% to 79% predicted and FEV1 / FVC < 0.7. For a diagnosis of moderate COPD, patients must have FEV1 40% to 59% predicted and FEV1 / FVC < 0.7.
3. Current or former smokers with > 20 pack-year smoking history.
4. Ability to provide informed consent.
5. Women subjects must be post-menopausal.

Exclusion Criteria:

1. Current or recent (within 4 weeks) acute exacerbation of chronic bronchitis
2. Current daily use of mineral or vitamin + mineral supplements or other natural health products that provide a daily dose of selenium that is greater than 100 µg
3. Current daily use of >5000 U of vitamin A, >1000 mg of vitamin C, or >800 U vitamin E
4. Known significant co-morbidity such as renal (creatinine > 150 mol/L) or hepatic disease (AST or ALT >3 times normal). Measurement of these will be a requirement of the study. Creatinine and Alanine aminotransferase (ALT) will be measured at the beginning and at the end of the study.
5. Known or suspected active cancer other than non-melanoma skin cancer.
6. Other concurrent major respiratory diagnosis other than COPD/asthma.
7. Plan to start statin drugs during the 12 weeks of study drug (may enroll if statins started >1 month before current study enrollment or deferred until study completion).
8. Consumption of brazil nuts.
9. Individuals who have homocystinuria
10. On niacin at a daily dose of 500 mg or higher for hyperlipidemia.
11. If you have allergies to products that contain dicalcium phosphate, talc sugarloaf, steric acid, or silica.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determine whether 12 weeks of selenium supplementation increases GPx-1 levels compared with placebo

SECONDARY OUTCOMES:
To determine whether selenium affects respiratory symptoms and function, and measures of inflammatory and infections markers.

CONTACTS AND LOCATIONS:
Overall Officials: Marek J Smieja, MD PhD FRCPC, Principal Investigator — Associate Professor, Dept. of Pathology & Molecular Medicine, McMaster University; Microbiologist & Infectious Disease Physician, Dept. of Laboratory Medicine
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada